CLINICAL TRIAL: NCT04741412
Title: SARS-CoV-2 Infections in Children and Adolescents: Course of COVID-19, Immune Responses, Complications and Long-term Consequences in Entire Households With Members Younger Than 18 Years
Brief Title: Pediatric SARS-CoV-2 Infections: Course of COVID-19, Immune Responses, Complications and Long-term Consequences
Acronym: PEDCOVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Holm Schneider, Head, Center of Ectodermal Dysplasias, University Hospital Erlangen
Other Study IDs: 212_20 B
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Hypohidrotic Ectodermal Dysplasia
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — serum, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypohidrotic Ectodermal Dysplasia: all household members with hypohidrotic ectodermal dysplasia (HED), a rare hereditary developmental disorder
- Control: individuals of the same age group, but without HED, including pregnant women

SUMMARY:
Longitudinal study of 56 households with at least one member who had COVID-19 to compare the course of illness, immune responses, and long-term consequences of SARS-CoV-2 infection in HED patients with those of control subjects of the same age group. Complete households are investigated, including women who are pregnant when exposed to the virus and their newborn child(ren).

ELIGIBILITY:
Inclusion Criteria:

* household with one or more members registered as patient(s) in the University Hospital Erlangen
* at least one person <18 years of age
* at least one household member who has or had a SARS-CoV-2 infection confirmed by a positive PCR test, detection of specific antibodies against this virus, or by development of COVID-19 symptoms after being in close contact with a person known to be infected with SARS-CoV-2
* informed consent

Exclusion Criteria:

* missing informed consent of one or more household members
* language barriers to communication that would prevent informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: households with children and/or adolescents and at least one member who has or had a SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
age-dependence of SARS-CoV-2 infection | 3 months from the point in time at which the first household member shows symptoms of COVID-19
  registry of household members with and without symptoms of COVID-19 (entire households)
percentage of household members infected by SARS-CoV-2 | 3 months from the point in time at which the first household member shows symptoms of COVID-19
  The infection rate is determined on the basis of specific PCR tests and detectibility of antibodies against SARS-CoV-2.
duration of primary COVID-19 symptoms | 2 months from the onset of COVID-19 symptoms
  The possible association between the length of time with symptoms of COVID-19 and specific immune responses, in particular the development of virus-neutralizing antibodies, is studied.
frequency of late-onset cardiovascular complications | 2-12 months from the onset of COVID-19 symptoms
  Patient-reported known and yet unknown long-term consequences of COVID-19 are registered and investigated further (questionnaire, specific data confirmed by clinical examination).
frequency of postviral fatigue | 2-12 months from the onset of COVID-19 symptoms
  Patient-reported symptoms of fatigue are registered (questionnaire).
frequency of noticeable temporary hair loss after COVID-19 | 2-12 months from the onset of COVID-19 symptoms
  Patient-reported extent of hair loss is registered (questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Holm Schneider, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Germany